CLINICAL TRIAL: NCT00989014
Title: Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled, Dose-Finding Study Investigating the Pharmacodynamics and Safety of Three Concentrations of CD07805/47 Topical Gel (0.07%, 0.18%, and 0.50%), Applied in Subjects With Moderate to Severe Erythematotelangiectatic Rosacea
Brief Title: Dose-Finding Study of CD07805/47 Topical Gel in Subjects With Erythematotelangiectatic Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18144
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2013-09

CONDITIONS: Erythematotelangiectatic Rosacea
Keywords: Erythematotelangiectatic; Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CD07805/47 0.5% Topical Gel (Experimental): 0.5% Topical Gel
  Interventions: Drug: CD07805/47
- CD07805/47 0.18% Topical Gel (Experimental): 0.18% Topical Gel
  Interventions: Drug: CD07805/47
- CD07805/47 0.07% Topical Gel (Experimental): 0.07% Topical Gel
  Interventions: Drug: CD07805/47
- CD07805/47 Vehicle Topical Gel (Placebo Comparator): Vehicle Topical Gel
  Interventions: Drug: CD07805/47 placebo

INTERVENTIONS:
Drug: CD07805/47 — 0.5% Topical Gel
  Arms: CD07805/47 0.5% Topical Gel
Drug: CD07805/47 — 0.18% Topical Gel
  Arms: CD07805/47 0.18% Topical Gel
Drug: CD07805/47 — 0.07% Topical Gel
  Arms: CD07805/47 0.07% Topical Gel
Drug: CD07805/47 placebo — Vehicle Topical Gel
  Arms: CD07805/47 Vehicle Topical Gel

SUMMARY:
This is a randomized, double-blind, parallel-group, vehicle-controlled, dose-finding study to investigate the pharmacodynamics and the safety of three dosages of CD07805/47 topical gel (0.07%, 0.18%, and 0.50%), after a single application in subjects with a clinical diagnosis of stable moderate to severe erythematotelangiectatic rosacea. Subjects will be randomized in a 1:1:1:1 ratio to receive either one of three CD07805/47 topical gel concentrations (0.07%, 0.18%, or 0.50%) or Vehicle Gel. All subjects will be treated with a single application (once daily dosing for one day) of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who is at least 18 years of age.
* Clinical diagnosis of stable moderate to severe erythematotelangiectatic rosacea.
* CEA (clinician's erythema assessment) score greater than or equal to 3 at Screening and on Treatment visit at baseline.
* PSA (patient self assessment) score of greater than or equal to 3 at Screening and on Treatment visit at baseline.
* Presence of 2 or fewer inflammatory facial lesions.

Exclusion Criteria:

* History of Raynaud's Syndrome, glaucoma, orthostatic hypotension, thromboangiitis obliterans, cerebral or coronary insufficiency, or depression.
* History of refractive surgery such as photorefractive keratectomy.
* The subject is being treated with monoamine oxidase (MAO) inhibitor, anti-depressants, barbiturates, opiates, sedatives, systemic anesthetics, alpha-agonists, beta blockers, antihypertensive agents, cardiac glycosides, or systemic anticoagulants.
* The subject is currently enrolled in an investigational drug or device study or participated in such a study in the past 3 months prior to enrollment and is still in the exclusion period on the day of the Treatment visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (5):
- United States (5):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Philadephia Institute of Dermatology, Fort Washington, Pennsylvania
  - Derm Research, Inc, Austin, Texas
  - J&S Studies, College Station, Texas
  - The Education & Research Foundation, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CD07805/47 0.5% Topical Gel | CD07805/47 0.18% Topical Gel | CD07805/47 0.07% Topical Gel | CD07805/47 Vehicle Topical Gel
Started | 31 | 31 | 28 | 32
Completed | 31 | 31 | 28 | 32
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD07805/47 0.5% Topical Gel | CD07805/47 0.18% Topical Gel | CD07805/47 0.07% Topical Gel | CD07805/47 Vehicle Topical Gel | Total
Number analyzed (Participants) | 31 | 31 | 28 | 32 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 27 | 29 | 117
  >=65 years | 0 | 1 | 1 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (11.87) | 46.3 (12.37) | 43.7 (10.74) | 46.7 (13.35) | 45.7 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 22 | 24 | 92
  Male | 6 | 10 | 6 | 8 | 30
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 28 | 32 | 122

OUTCOME MEASURES:

1. Primary Outcome: Response Rate for Achieving a 2 Grade Improvement on Clinician's Erythema Assessment (CEA) and Patient Self Assessment (PSA) Over 12 Hours After Dosing.
Time Frame: Baseline and every hour for 12 hours following application
Measure: Number; unit: participants
Arm/Group | CD07805/47 0.5% Topical Gel | CD07805/47 0.18% Topical Gel | CD07805/47 0.07% Topical Gel | CD07805/47 Vehicle Topical Gel
Number analyzed (Participants) | 31 | 31 | 28 | 32
participants | 17 | 10 | 7 | 4

ADVERSE EVENTS:
Arm/Group | CD07805/47 0.5% Topical Gel | CD07805/47 0.18% Topical Gel | CD07805/47 0.07% Topical Gel | CD07805/47 Vehicle Topical Gel
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 4/31 | 1/31 | 3/28 | 5/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD07805/47 0.5% Topical Gel (N=31) | CD07805/47 0.18% Topical Gel (N=31) | CD07805/47 0.07% Topical Gel (N=28) | CD07805/47 Vehicle Topical Gel (N=32)
Headache (Nervous system disorders) | 3 | 0 | 0 | 2
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days